CLINICAL TRIAL: NCT01767350
Title: Study Aimed at Determining the Relation Between the Administered Dose and Exposure to Immunosuppressive Medication in Children After Solid Organ Transplantation
Brief Title: Determinants of Immunosuppressive Dose Requirements in Children After Solid Organ Transplantation
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Noël Knops, Dr, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S55088
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Transplantation Infection
Keywords: Pediatric transplantation; Pharmacogenetics; Pharmacokinetics; Calcineurin inhibitors; CYP3A; Pgp
MeSH Terms: interventions — DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tube of whole blood (8 ml) to be processed for DNA extraction and storage
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- children with organ transplant: Subjects who received an solid organ transplant at our institution at the age of 0-19 yrs and who were subject to pharmacokinetic evaluation during their follow up. Additional blood withdrawal for DNA will be performed
  Interventions: Procedure: Blood withdrawal for DNA

INTERVENTIONS:
Procedure: Blood withdrawal for DNA — Single withdrawal of 8 ml whole blood for DNA analysis, during a "standard" blood collection as part of standard clinical follow up.
  Other Names: not applicalble

SUMMARY:
The long-term success of solid organ transplantation is largely dependent on the efficacy of immunosuppressive medication. Unfortunately, for the most important agents the correct drug levels are difficult to attain, with potential severe consequences of drug under- or overexposure. In addition there is a large variation in dose requirements within and between different subjects. Clinical studies have demonstrated that a better control of drug exposure can improve outcome. A large set of patient characteristics appear important in determining dose requirements in adults, in particular genetic variation in genes involved in drug metabolism. In children relative dose requirements are increased compared to adults, but is not known why and the role of pharmacogenetic variation has not been described.

Our study aims to describe relative dose requirements in children after solid organ transplantation with the help of clinical and laboratory data obtained during regular hospital visits (retrospective). In addition we will assess their genotype for genes involved in the metabolism of immunosuppressives.

DETAILED DESCRIPTION:
The success of solid organ transplantation is for an important part determined by the potency of the immunosuppressive regime to prevent allograft rejection. Depending on the type of organ transplanted current 5-year graft survival for liver is circa 70% and for kidney almost 80% (1-3). Although acute rejection has become less a problem, analyses of data on the follow-up of solid organ recipients has demonstrated that long-term allograft survival has not improved much in the last decade. The life expectancy of a donor organ appears limited due to phenomena such as chronic, antibody mediated, rejection and the toxic effects of immunosuppressive medication.

Unfortunately, the most commonly applied immunosuppressive agents (in particular the calcineurin-inhibitors) possess a narrow therapeutic index with potential severe consequences of drug under- or overexposure. Furthermore, in clinical practice optimal dosing is difficult to achieve due to important inter- and intraindividual variation in drug pharmacokinetics. Consequently attention has shifted towards designing a "tailored immunosuppressive maintenance therapy", aimed at optimization of drug efficacy and the prevention of these unintended and possible deleterious side effects in the individual recipient. For a "perfect fit" this entails a fundamental knowledge of the individual characteristics of the recipient and its graft in relation to the pharmacodynamic and -kinetic properties of the agent.

A complex and often interdependent set of factors appears relevant in determining drug exposure. These include recipient characteristics such as age, race, body composition, organ function (intestine-liver-kidney), food and concomitant medication intake, but also graft-related characteristics such as: seize, donor-age, and time after transplantation. Longitudinal and cross-sectional analysis of clinical and genetic co-variables in allograft recipient cohorts has identified several single nucleotide polymorphisms (SNPs) in genes encoding for enzymes and transporters involved in drug metabolism(CYP3A4, CYP3A5, MDR1), which were associated with differences in dosing and toxicity (4-10). In particular carriers of a common polymorphism in CYP3A5 (designated CYP3A5*1) demonstrate a 25-40% increase in tacrolimus clearance and a 2-3 fold increase in dose requirements.

In children the dose requirements per kg bodyweight to attain desired blood concentrations are approximately 2.7 fold higher for patients under 5 years and 1.9 fold higher for patients aged 5 to 12 years when compared to older patients11-14. Age-related differences in expression of enzymes or transporters involved in drug metabolism might play an important role. Fakhoury et al demonstrated an increase in intestinal CYP3A4/5 mRNA and protein expression from childhood to adulthood (15). In addition other factors such as intestinal transit time and length, body composition, protein binding, body metabolism and organ function, might be important in determining dose requirements in children (16-18). The importance of the aforementioned genetic polymorphisms on long-term dose requirements have not been studied in children.

Objective:

To describe dose requirements of immunosuppressive medication in relation to a set of clinical and non-clinical (genetic) factors in a cohort of pediatric recipients of a solid organ allograft.

Methods:

A retrospective study in a single center (University Hospitals Leuven) with an active program for pediatric kidney, liver and intestinal transplantation. The study population consists of subjects who received a solid organ transplant (liver, kidney, intestine, combined) between 0 and 18 years of age.

As a part of their standard care patients are admitted to the department for a yearly check-up after transplantation. During this admission a set of investigations are performed to evaluate the current medical situation, including an elaborate pharmacokinetic (PK) assessment. Patient characteristics and clinical data (age, bodyweight, sex, type of graft, cause of organ failure, co-medication, laboratory results, PK data) will be retrieved from the patient files concerning these follow-up admissions. In addition patients and/or their parents will be requested permission to collect one extra tube of whole blood (ca 8 ml) for DNA analysis during a standard blood collection at a regular hospital/outpatient visit.

After collection patient data will be given a code for further anonymous storage and analysis. DNA SNP analysis will take place at our laboratory for pediatric nephrology with PCR.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric recipients of a solid organ transplantation in our hospital
* Extensive pharmacokinetic study of immunosuppression (AUC) performed during follow up
* Consent of child/caretaker

Exclusion Criteria:

-

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric recipients of a solid organ transplantation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Relative dose requirement of tacrolimus, ciclosporin or MMF | 1 yr
  analysis of retrospective data concerning pharmacokinetic assessment as part of standard clinical care

SECONDARY OUTCOMES:
Pharmacogenetic genotype | 1 yr
  Analysis of DNA obtained during a regular hospital visit for genetic variants relevant for metabolism of immunosuppression according to literature (CYP3A4, CYP3A5, MDR1, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Noel Knops, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Background] Cai J, Terasaki PI. Induction immunosuppression improves long-term graft and patient outcome in organ transplantation: an analysis of United Network for Organ Sharing registry data. Transplantation. 2010 Dec 27;90(12):1511-5. doi: 10.1097/TP.0b013e3181fecfcb. PMID 21057388
- [Background] Opelz G, Susal C, Ruhenstroth A, Dohler B. Impact of HLA compatibility on lung transplant survival and evidence for an HLA restriction phenomenon: a collaborative transplant study report. Transplantation. 2010 Oct 27;90(8):912-7. doi: 10.1097/TP.0b013e3181f2c981. PMID 20808265
- [Background] Opelz G, Dohler B; Collaborative Transplant Study. Influence of immunosuppressive regimens on graft survival and secondary outcomes after kidney transplantation. Transplantation. 2009 Mar 27;87(6):795-802. doi: 10.1097/TP.0b013e318199c1c7. PMID 19300179
- [Background] Staatz CE, Goodman LK, Tett SE. Effect of CYP3A and ABCB1 single nucleotide polymorphisms on the pharmacokinetics and pharmacodynamics of calcineurin inhibitors: Part I. Clin Pharmacokinet. 2010 Mar;49(3):141-75. doi: 10.2165/11317350-000000000-00000. PMID 20170205
- [Background] Staatz CE, Goodman LK, Tett SE. Effect of CYP3A and ABCB1 single nucleotide polymorphisms on the pharmacokinetics and pharmacodynamics of calcineurin inhibitors: Part II. Clin Pharmacokinet. 2010 Apr;49(4):207-21. doi: 10.2165/11317550-000000000-00000. PMID 20214406
- [Background] de Jonge H, Kuypers DR. Pharmacogenetics in solid organ transplantation: current status and future directions. Transplant Rev (Orlando). 2008 Jan;22(1):6-20. doi: 10.1016/j.trre.2007.09.002. PMID 18631854
- [Background] de Jonge H, Naesens M, Kuypers DR. New insights into the pharmacokinetics and pharmacodynamics of the calcineurin inhibitors and mycophenolic acid: possible consequences for therapeutic drug monitoring in solid organ transplantation. Ther Drug Monit. 2009 Aug;31(4):416-35. doi: 10.1097/FTD.0b013e3181aa36cd. PMID 19536049
- [Background] Zhou SF, Di YM, Chan E, Du YM, Chow VD, Xue CC, Lai X, Wang JC, Li CG, Tian M, Duan W. Clinical pharmacogenetics and potential application in personalized medicine. Curr Drug Metab. 2008 Oct;9(8):738-84. doi: 10.2174/138920008786049302. PMID 18855611
- [Background] Rosso Felipe C, de Sandes TV, Sampaio EL, Park SI, Silva HT Jr, Medina Pestana JO. Clinical impact of polymorphisms of transport proteins and enzymes involved in the metabolism of immunosuppressive drugs. Transplant Proc. 2009 Jun;41(5):1441-55. doi: 10.1016/j.transproceed.2009.03.024. PMID 19545654
- [Background] Claeys T, Van Dyck M, Van Damme-Lombaerts R. Pharmacokinetics of tacrolimus in stable paediatric renal transplant recipients. Pediatr Nephrol. 2010 Feb;25(2):335-42. doi: 10.1007/s00467-009-1331-6. Epub 2009 Nov 3. PMID 19885684
- [Background] Montini G, Ujka F, Varagnolo C, Ghio L, Ginevri F, Murer L, Thafam BS, Carasi C, Zacchello G, Plebani M. The pharmacokinetics and immunosuppressive response of tacrolimus in paediatric renal transplant recipients. Pediatr Nephrol. 2006 May;21(5):719-24. doi: 10.1007/s00467-006-0014-9. Epub 2006 Mar 21. PMID 16550361
- [Background] Naesens M, Salvatierra O, Li L, Kambham N, Concepcion W, Sarwal M. Maturation of dose-corrected tacrolimus predose trough levels in pediatric kidney allograft recipients. Transplantation. 2008 Apr 27;85(8):1139-45. doi: 10.1097/TP.0b013e31816b431a. PMID 18431234
- [Background] Ferraris JR, Argibay PF, Costa L, Jimenez G, Coccia PA, Ghezzi LF, Ferraris V, Belloso WH, Redal MA, Larriba JM. Influence of CYP3A5 polymorphism on tacrolimus maintenance doses and serum levels after renal transplantation: age dependency and pharmacological interaction with steroids. Pediatr Transplant. 2011 Aug;15(5):525-32. doi: 10.1111/j.1399-3046.2011.01513.x. Epub 2011 Jun 28. PMID 21711429
- [Background] Fakhoury M, Litalien C, Medard Y, Cave H, Ezzahir N, Peuchmaur M, Jacqz-Aigrain E. Localization and mRNA expression of CYP3A and P-glycoprotein in human duodenum as a function of age. Drug Metab Dispos. 2005 Nov;33(11):1603-7. doi: 10.1124/dmd.105.005611. Epub 2005 Jul 27. PMID 16049125
- [Background] Kanamori M, Takahashi H, Echizen H. Developmental changes in the liver weight- and body weight-normalized clearance of theophylline, phenytoin and cyclosporine in children. Int J Clin Pharmacol Ther. 2002 Nov;40(11):485-92. doi: 10.5414/cpp40485. PMID 12698985
- [Background] Kearns GL, Abdel-Rahman SM, Alander SW, Blowey DL, Leeder JS, Kauffman RE. Developmental pharmacology--drug disposition, action, and therapy in infants and children. N Engl J Med. 2003 Sep 18;349(12):1157-67. doi: 10.1056/NEJMra035092. No abstract available. PMID 13679531
- [Background] Bartelink IH, Rademaker CM, Schobben AF, van den Anker JN. Guidelines on paediatric dosing on the basis of developmental physiology and pharmacokinetic considerations. Clin Pharmacokinet. 2006;45(11):1077-97. doi: 10.2165/00003088-200645110-00003. PMID 17048973